CLINICAL TRIAL: NCT01663623
Title: A Phase 3, Multi-Center, Multinational, Randomized, Double-Blind, Study to Evaluate the Efficacy and Safety of Belimumab (HGS1006) in Combination With Azathioprine for the Maintenance of Remission in Wegener's Granulomatosis and Microscopic Polyangiitis
Brief Title: Belimumab in Remission of VASculitis
Acronym: BREVAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Human Genome Sciences Inc., a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115466
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Vasculitis
Keywords: Wegener's Granulomatosis; anti-MPO; WG; Belimumab; GPA; anti-proteinase 3; anti-neutrophil cytoplasmic antibody; anti-myeloperoxidase; Granulomatosis with polyangiitis; Vasculitis; Autoimmune Diseases; Microscopic Polyangiitis; anti-PR3; ANCA; MPA; Systemic Vasculitis
MeSH Terms: conditions — Vasculitis; Granulomatosis with Polyangiitis; Autoimmune Diseases; Microscopic Polyangiitis; Systemic Vasculitis | interventions — belimumab; Azathioprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo plus azathioprine (Placebo Comparator): Placebo IV plus oral azathioprine 2 mg/kg/day; placebo administered on Days 0, 14, 28, and then every 28 days until the end of the study. If the results in the double-blind period show that belimumab is safe and effective, then participants have the option to receive treatment with belimumab in a 6-month open-label extension phase. Placebo patients who opt to participate in the extension will receive belimumab 10 mg/kg IV every 28 days plus oral azathioprine 2 mg/kg/day for an additional 6 months.
  Interventions: Biological: Placebo; Drug: Azathioprine
- Belimumab 10 mg/kg plus azathioprine (Experimental): Belimumab 10 mg/kg IV plus oral azathioprine 2 mg/kg/day; belimumab administered on Days 0, 14, 28, and then every 28 days until the end of the study. If the results in the double-blind period show that belimumab is safe and effective, then participants have the option to continue treatment with belimumab in a 6-month open-label extension phase. Patients who opt to participate in the extension will continue to receive belimumab 10 mg/kg IV every 28 plus oral azathioprine 2 mg/kg/day days for an additional 6 months.
  Interventions: Biological: Belimumab 10 mg/kg; Drug: Azathioprine

INTERVENTIONS:
Biological: Placebo — Placebo
  Arms: Placebo plus azathioprine
Biological: Belimumab 10 mg/kg — Belimumab 10 mg/kg
  Other Names: BENLYSTA™
  Arms: Belimumab 10 mg/kg plus azathioprine
Drug: Azathioprine — Azathioprine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of belimumab, in combination with azathioprine, for the maintenance of remission following a standard induction regimen in patients with Wegener's granulomatosis or microscopic polyangiitis. The random assignment in this study is "1 to 1" which means that participants have an equal chance of receiving belimumab or placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis Wegener's granulomatosis or microscopic polyangiitis by Chapel Hill criteria.
* Disease flare in the past 26 weeks requiring treatment with high dose corticosteroids and 1 of the following medications: rituximab, oral cyclophosphamide OR IV cyclophosphamide.
* Tested positive for anti-proteinase 3 (anti-PR3) or anti-myeloperoxidase (anti-MPO) antibodies at any time prior to enrollment.
* Achieve remission no more than 26 weeks after first dose of induction treatment. Remission is defined as a Birmingham Vasculitis Activity (BVAS) score of 0 and receiving less than 10 mg/day of oral prednisone (or equivalent) on 2 consecutive visits 21 to 35 days apart.
* Maintenance therapy on this study must start no more than 2 weeks after confirmation of remission.

Key Exclusion Criteria:

* Pregnant or nursing.
* Receipt of a B cell targeted therapy (other than rituximab) at anytime
* Receipt of an investigational biological agent within the past 60 days.
* Required management of acute or chronic infections within the past 60 days.
* Current drug or alcohol abuse or dependence.
* Current or past positive test for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* History of severe allergic reaction to contrast agents or biological medicines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (77):
- United States (21):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Covina, California
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, San Leandro, California
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, West Springfield, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, Milwaukee, Wisconsin
- Australia (4):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, New Lambton, New South Wales
  - GSK Investigational Site, Malvern, Victoria
  - GSK Investigational Site, Liverpool
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
- Canada (3):
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Prague, Czechia
- France (4):
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Rennes
- Germany (8):
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Kirchheim unter Teck
  - GSK Investigational Site, München
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
- GSK Investigational Site, Dublin, Ireland
- Italy (6):
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Torrette Di Ancona, The Marches
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Reggio Emilia
- GSK Investigational Site, México, Mexico
- Norway (2):
  - GSK Investigational Site, Kristiansand
  - GSK Investigational Site, Oslo
- Peru (2):
  - GSK Investigational Site, Callao
  - GSK Investigational Site, Lima
- Poland (4):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lublin
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Stavropol
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
- GSK Investigational Site, Stockholm, Sweden
- Switzerland (3):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Sankt Gallen
  - GSK Investigational Site, Zurich
- United Kingdom (5):
  - GSK Investigational Site, Reading, Berkshire
  - GSK Investigational Site, Aberdeen
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London
  - GSK Investigational Site, Oxford

REFERENCES:
- [Derived] Jayne D, Blockmans D, Luqmani R, Moiseev S, Ji B, Green Y, Hall L, Roth D, Henderson RB, Merkel PA; BREVAS Study Collaborators. Efficacy and Safety of Belimumab and Azathioprine for Maintenance of Remission in Antineutrophil Cytoplasmic Antibody-Associated Vasculitis: A Randomized Controlled Study. Arthritis Rheumatol. 2019 Jun;71(6):952-963. doi: 10.1002/art.40802. Epub 2019 Apr 16. PMID 30666823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with diagnosis of Granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA) were randomized in this study. The study was conducted at 37 centers in 15 countries in North America, Central America, South America, Western Europe, Eastern Europe, and Australia during 20 March 2013 - 06 February 2017.
Pre-assignment Details: A total of 164 participants were screened and 106 were enrolled and randomized in a 1:1 ratio to receive placebo or belimumab 10 milligram per kilogram (mg/kg). Of which, 105 received at least 1 dose of study agent and one participant was randomized in error.
Groups:
- Placebo: Participants were administered induction therapy (corticosteroids and either cyclophosphamide or rituximab) in the 6 months leading up to randomization. After randomization, participants were administered matching placebo intravenously over 1 hour, at Day 0, 14, 28 and every 28 days thereafter until 12 months after the last subject was randomized. All participants received oral azathioprine at a target dose of 2 milligram per kilogram per day (mg/kg/day). In Belgium-only open-label extension, all participants received belimumab 10mg/day every 28 days until Week 24, with a final evaluation at Week 28.
- Belimumab 10 mg/kg: Participants were administered induction therapy (corticosteroids and either cyclophosphamide or rituximab) in the 6 months leading up to randomization. After randomization, participants were administered belimumab 10 mg/kg intravenously over 1 hour, at Day 0, 14, 28 and every 28 days thereafter until 12 months after the last subject was randomized. All participants received oral azathioprine at a target dose of 2 mg/kg/day. In Belgium-only open-label extension, all participants received belimumab 10 mg/kg every 28 days until Week 24, with a final evaluation at Week 28.
Period: Overall Study
Arm/Group | Placebo | Belimumab 10 mg/kg
Started | 52 | 53
Completed | 40 | 33
Not Completed | 12 | 20
Not completed — Adverse Event | 3 | 7
Not completed — Lack of Efficacy | 5 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — Other-Study closed/terminated | 1 | 1
Not completed — Physician Decision | 1 | 4
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Belimumab 10 mg/kg | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (13.56) | 56.2 (13.59) | 54.8 (13.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 27 | 27 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 1 | 1 | 2
  American Indian or Alaskan Native | 5 | 6 | 11
  Central/South Asian Heritage | 2 | 0 | 2
  White | 44 | 46 | 90

OUTCOME MEASURES:

1. Primary Outcome: Time to First Relapse
Description: Time to relapse is defined as the number of days from Day 0 until the participant experienced a relapse (relapse date - treatment start date +1). Only post-baseline relapses were considered in these analyses. Only relapses occurring up to and including the last visit date in the double-blind treatment period were considered in these analyses. Intent-to-treat population comprised of all randomized participants who received at least one dose of study agent (belimumab or placebo). NA indicates that the data was not available as the Number of events is too low to estimate the value. Median and Inter-quartile range were presented and were based on Kaplan Meier estimates.
Time Frame: Approximately up to 4 years
Population: Intent-to-treat population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 52 | 53
Days | NA [789.0 to NA] — Kaplan Meier statistics could not be estimated where the number of events is too low. Hence it is NA. | NA [NA to NA] — Kaplan Meier statistics could not be estimated where the number of events is too low. Hence it is NA.
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; p = 0.884, Cox Proportional Hazards model — Cox proportional Hazards (Wald Chi Square); Analysis was adjusted for ANCA type, disease stage at induction and induction regimen; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.44 to 2.59] — Analysis performed using a Cox Proportional Hazards model with covariates treatment group, Actual ANCA type, Actual disease stage at induction and Actual induction regimen

2. Secondary Outcome: Number of Participants With Major Relapse During the Double-blind Phase of the Study
Description: Data for number of participants with major relapse [defined as experiencing at least 1 major Birmingham Vasculitis Activity Score (BVAS) item] during the double-bind phase of the study was reported. Analysis was performed using a Cox proportional hazard model.
Time Frame: Approximately up to 4 years
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 52 | 53
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the start of study agent administration (Day 0) through 8 weeks following administration of the last dose of study agent (approximately up to 4 years).
Description: Intent to treat population. Participants who discontinued treatment, all AE were collected through 8 weeks following the last dose of study agent. All SAEs were collected until relapse or the study was analyzed for the primary endpoint and study sites are informed that SAE data collection can cease, whichever occurs first.
Arm/Group | Placebo | Belimumab 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/52 | 1/53
Serious Adverse Events (participants affected / at risk) | 16/52 | 18/53
Other Adverse Events (participants affected / at risk) | 33/52 | 32/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | Belimumab 10 mg/kg (N=53)
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 2
Anaphylactic reaction (Immune system disorders) | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Idiopathic orbital inflammation (Eye disorders) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | Belimumab 10 mg/kg (N=53)
Nasopharyngitis (Infections and infestations) | 10 | 6
Upper respiratory tract infection (Infections and infestations) | 8 | 7
Urinary tract infection (Infections and infestations) | 4 | 5
Bronchitis (Infections and infestations) | 6 | 1
Influenza (Infections and infestations) | 1 | 5
Gastroenteritis (Infections and infestations) | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 2
Fatigue (General disorders) | 7 | 7
Pyrexia (General disorders) | 2 | 6
Headache (Nervous system disorders) | 7 | 5
Rash (Skin and subcutaneous tissue disorders) | 3 | 5
Hypertension (Vascular disorders) | 4 | 3

LIMITATIONS AND CAVEATS:
The sample size was small as it was truncated from approximately 300 to 100 participants, largely owing to a change in standard of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-02-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT01663623/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT01663623/SAP_001.pdf